CLINICAL TRIAL: NCT02858154
Title: Comparison of High Flow Nasal Cannula Therapy to Nasal Oxygen (O2) as a Treatment for Obstructive Sleep Apnea (OSA) in Infants
Brief Title: Comparison of High Flow Nasal Cannula Therapy to Nasal Oxygen as a Treatment for Obstructive Sleep Apnea in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Neepa Gurbani, DO, DO, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN001-HFNC and OSA
Record Dates: First submitted 2016-07-25; First posted 2016-08-08 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; obstructive sleep apnea; infants; high flow nasal cannula; HFNC
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HFNC and low flow oxygen by nasal cannula (Other): All subjects will receive 3-4 hours of experimental treatment (HFNC) during a research portion of a PSG and then for the 6-8 hours of clinically ordered PSG will receive active comparator (low flow oxygen by nasal cannula)
  Interventions: Other: HFNC; Other: Low flow oxygen by nasal cannula

INTERVENTIONS:
Other: HFNC — All subjects will have a 3-4 hour intervention of HFNC to test effectiveness and safety for treating OSA
  Other Names: High Flow Nasal Cannula
Other: Low flow oxygen by nasal cannula — All subjects will have a 6 to 8 hours intervention during the clinically scheduled PSG of titration of oxygen by nasal cannula (standard of care) to manage sleep apnea

SUMMARY:
This is a small pilot study that will compare High Flow Nasal Cannula (HFNC) therapy to oxygen nasal cannula therapy on infants who have obstructive sleep apnea (OSA) and are scheduled for a clinically ordered sleep study called polysomnography (PSG). The HFNC procedure uses humidified room air delivered by nasal cannula at higher pressures and will test if HFNC can control OSA in infants better or as well as low flow nasal oxygen, the current clinical standard of care. All the infants in the study will have a brief test period of about 3 to 4 hours with the HFNC before participants begin their standard clinical PSG for titration of oxygen by nasal cannula for treatment of OSA.

DETAILED DESCRIPTION:
The current standard of care for treating OSA in infants less than 6 months and frequently up to 12 months of age is with a continuous flow of oxygen by nasal cannula. This is generally referred to as nasal continuous positive airway pressure or NCPAP. A nasal cannula is used with oxygen at low flows of between 1/4 to 1 liter per minute (l/m) to deliver supplemental oxygen to reduce oxygen desaturations associated with apneic episodes and to provide a positive pressure flow to maintain an open airway.

High Flow Nasal Cannula (HFNC) therapy is a non-invasive treatment providing respiratory support. In this study, HFNC is designed to administer a heated and humidified mixture of air at a flow higher than the patient's inspiratory flow. There is currently no single, simple definition of high flow. In infants, it usually refers to a flow of >2 l/min and in children it is considered >6 l/min. High flow presents several advantages over conventional 'low-flow' oxygen therapy in terms of humidification, oxygenation, gas exchange, and breathing pattern. Several studies have shown that a flow higher than the patient's inspiratory flow provides better oxygen delivery than low-flow oxygen therapy or high-concentration oxygenation mask. This observation has been explained as the effect of a high flow on the oropharyngeal dead space, washing out oxygen depleted gas and reducing carbon dioxide (CO2) rebreathing. The extrathoracic dead space is proportionally two to three times greater in children than in adults. It may measure up to 3 mL/kg in newborns and becomes similar to the adult volume only after 6 years of age (0.8 mL/kg). Consequently, the younger a child is, the greater the effect of a high flow on oxygenation and CO2 clearance.

This pilot study is to compare standard of care low flow nasal oxygen to the effectiveness of HFNC therapy in infants aged 12 months and younger to treat OSA. The study intervention will occur for approximately 3 to 4 hours immediately prior to a scheduled clinical PSG. Subjects will be prepared for standard clinical PSG and after asleep, the intervention will be titration of room air at different pressure flows delivered by a HFNC system. At the end of the research portion of the PSG, the clinical PSG will begin with the standard of care treatment, the nasal oxygen titration for OSA. The results of the clinical PSG will serve as control comparison for the research intervention.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤ 12 months
* Diagnosis of OSA from previous PSG

Exclusion Criteria:

* Infants who on previous PSG had central apneas > 50% of the AHI

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2016-02; Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neepa Gurbani, DO, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Zarmina Ehsan, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (2):
- United States (2):
  - Children's Mercy Hospital, Kansas City, Kansas
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sreenan C, Lemke RP, Hudson-Mason A, Osiovich H. High-flow nasal cannulae in the management of apnea of prematurity: a comparison with conventional nasal continuous positive airway pressure. Pediatrics. 2001 May;107(5):1081-3. doi: 10.1542/peds.107.5.1081. PMID 11331690
- [Background] Kotecha SJ, Adappa R, Gupta N, Watkins WJ, Kotecha S, Chakraborty M. Safety and Efficacy of High-Flow Nasal Cannula Therapy in Preterm Infants: A Meta-analysis. Pediatrics. 2015 Sep;136(3):542-53. doi: 10.1542/peds.2015-0738. Epub 2015 Aug 17. PMID 26283781
- [Background] Milesi C, Boubal M, Jacquot A, Baleine J, Durand S, Odena MP, Cambonie G. High-flow nasal cannula: recommendations for daily practice in pediatrics. Ann Intensive Care. 2014 Sep 30;4:29. doi: 10.1186/s13613-014-0029-5. eCollection 2014. PMID 25593745

RESULTS

PARTICIPANT FLOW:
Groups:
- HFNC Followed by Clinically Ordered Low Flow Oxygen Via Nasal Cannula: All subjects received HFNC followed by clinically ordered low flow oxygen via nasal cannula.
  HFNC: All subjects will have a 3-4 hour intervention of HFNC to test effectiveness and safety for treating OSA
  Low flow oxygen by nasal cannula: All subjects will have a 6 to 8 hours intervention during the clinically scheduled PSG of titration of oxygen by nasal cannula (standard of care in infants) to control sleep apnea and desaturations
Period: HFNC 3-4 Hours
Arm/Group | HFNC Followed by Clinically Ordered Low Flow Oxygen Via Nasal Cannula
Started | 9
Completed | 9
Not Completed | 0
Period: Clinically Ordered PSG/Low Flow Oxygen
Arm/Group | HFNC Followed by Clinically Ordered Low Flow Oxygen Via Nasal Cannula
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Children With OSA Receiving HFNC and Low Flow Oxygen With Nasal Cannula: All subjects will receive 3-4 hours of experimental treatment (HFNC) during a research portion of a PSG and then for the 6-8 hours of clinically ordered PSG will receive active comparator (oxygen by nasal cannula)
  HFNC: All subjects will have a 3-4 hour intervention of HFNC to test effectiveness and safety for treating OSA
  Oxygen by Cannula: All subjects will have a 6 to 8 hours intervention during the clinically scheduled PSG of titration of oxygen by nasal cannula (standard of care) to control sleep apnea and desaturations
Arm/Group | Children With OSA Receiving HFNC and Low Flow Oxygen With Nasal Cannula
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 1.33 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Average AHI Diagnostic Sleep Study Compared to Average AHI With Improvement in OSA With HFNC
Description: AHI will be compared from diagnostic sleep study to average AHI with improvement in OSA with HFNC
Time Frame: End of visit (12 hours)
Population: We analyzed subjects who had improvement in AHI with HFNC compared to the diagnostic study.
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- Average AHI Diagnostic Sleep Study Compared to Average AHI With Improvement in OSA With HFNC: All subjects will receive 3-4 hours of experimental treatment (HFNC) during a research portion of a PSG and then for the 6-8 hours of clinically ordered PSG will receive low flow oxygen by nasal cannula.
Arm/Group | Average AHI Diagnostic Sleep Study Compared to Average AHI With Improvement in OSA With HFNC
Number analyzed (Participants) | 4
events/hour
  AHI on diagnostic study | 15.6 (5.65)
  AHI with improvement in OSA with HFNC | 5.12 (2.5)

2. Primary Outcome: AHI From Diagnostic Sleep Study Compared to AHI From Sleep Study Improvement in OSA With Low Flow Oxygen Via Nasal Cannula
Description: All subjects will receive 3-4 hours of experimental treatment (HFNC) during a research portion of a PSG and then for the 6-8 hours of clinically ordered PSG will receive low flow oxygen by nasal cannula.
Time Frame: end of visit (12 hours)
Population: Compared AHI with low flow oxygen via nasal cannula compared to diagnostic sleep study AHI.
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- Average AHI Diagnostic Study Compared to Average AHI With Improvement in OSA With Low Flow Oxygen: All subjects will receive 3-4 hours of experimental treatment (HFNC) during a research portion of a PSG and then for the 6-8 hours of clinically ordered PSG will receive low flow oxygen by nasal cannula.
Arm/Group | Average AHI Diagnostic Study Compared to Average AHI With Improvement in OSA With Low Flow Oxygen
Number analyzed (Participants) | 9
events/hour
  AHI from diagnostic sleep study | 13.44 (5.36)
  AHI from improvement in OSA with low flow oxygen by nasal cannula | 4.9 (3.12)

ADVERSE EVENTS:
Time Frame: 12 hours (duration of intervention)
Groups:
- HFNC for the First 3-4 Hours of the Study Followed by Clinically Ordered Low Flow Oxygen.: All subjects will receive 3-4 hours of experimental treatment (HFNC) during a research portion of a PSG and then 6-8 hours of clinically ordered PSG with low flow oxygen by nasal cannula for the remainder of the study. Since both interventions were done on the same night the sleep study with the first 3-4 hours of the sleep study with HFNC and the remainder 6-8 hours with clinically ordered PSG with low flow oxygen via nasal cannula the adverse events are reported for the duration of the study interventions.
Arm/Group | HFNC for the First 3-4 Hours of the Study Followed by Clinically Ordered Low Flow Oxygen.
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT02858154/Prot_SAP_000.pdf